CLINICAL TRIAL: NCT03851393
Title: Validation of Peptest™ for the Detection of Reflux in Cough; Induction of Cough in Healthy Volunteers
Brief Title: Validation of Peptest™ for the Detection of Reflux in Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Acadmed130514
Record Dates: First submitted 2014-05-15; First posted 2019-02-22 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cough
Keywords: Cough; Reflux; Pepsin; Peptest
MeSH Terms: conditions — Cough; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptest™ analysis of saliva pepsin (Experimental): Induction of cough with inhaled citric acid and measurement of saliva pepsin following citric acid cough challenge using the peptest lateral device
  Interventions: Other: Induction of cough with inhaled citric acid; Procedure: Peptest™ analysis of saliva pepsin; Diagnostic Test: Peptest™

INTERVENTIONS:
Other: Induction of cough with inhaled citric acid — perform artificially induced cough by inhalation of citric acid at various strengths
Procedure: Peptest™ analysis of saliva pepsin — collect patient saliva for analysis of pepsin levels
Diagnostic Test: Peptest™ — The Peptest™ lateral flow device

SUMMARY:
Chronic cough is a common presenting problem which has a significant impact on quality of life. Gastro-oesophageal reflux (GOR) is a common cause of chronic cough and reflux of stomach contents into the airways has been implicated in the pathogenesis of a number of respiratory diseases. Clinical history in patients with suspected reflux can aid in the diagnosis but traditional investigations for GOR including 24hr oesophageal pH monitoring or endoscopy are not reliable diagnostic tools since the reflux may be non acidic.

The detection of pepsin in the sputum, saliva or bronchial biopsy has been found to be an accurate marker of reflux into the airways. Pepsin is solely produced by parietal cells in the stomach. The presence of pepsin in the upper airways therefore indicates reflux. Studies have demonstrated that pepsin was frequently found in laryngeal biopsies and sputum of patients with signs and symptoms of airways reflux and that Nissen fundoplication resulted in a decrease in pepsin detection alongside an improvement in symptoms. The Peptest™ lateral flow device has been shown to be effective in the detection of pepsin in sputum and saliva of patients with chronic cough and gastro-oesophageal reflux. The investigators have detected pepsin in expectorated saliva during episodes of cough, apparently supporting a diagnosis of airways reflux. Critics, however, have suggested that the act coughing itself is responsible for the reflux.

This study aims to identify if cough induced by inhaled citric acid in healthy adult volunteers leads to detectable pepsin in expectorated saliva.

ELIGIBILITY:
Inclusion Criteria:

* A negative score for airway reflux (HARQ score <13).
* Provision of informed consent.

Exclusion Criteria:

* Participants with a positive score for airway reflux (HARQ score >13).
* Chronic respiratory disease.
* Acute gastro-respiratory illness at the time of the study.
* Participants who will be physically unable to undergo sputum collection or cough induction.
* Those who are unwilling to undergo cough challenge and induction of cough.
* Smoking or consumption of food, caffeinated or carbonated beverages for 30 minutes prior to sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
level of pepsin in saliva following a citric acid cough challenge | 3 months
  detecting the levels of pepsin in saliva following Citric acid induced cough

SECONDARY OUTCOMES:
normal range of saliva pepsin | 3 months
  record normal range of saliva pepsin following citric acid cough challenge

CONTACTS AND LOCATIONS:
Overall Officials: Alyn Morice, MD, FRCP, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull Clinical Trials Unit, Respiratory academic department, Cottingham, Yorkshire, United Kingdom

REFERENCES:
- See also: Publication Link — https://thorax.bmj.com/content/68/Suppl_3/A19.2